CLINICAL TRIAL: NCT06566924
Title: The Effect of Standardised Patient Simulation on Nursing Students' Knowledge, Skills and Satisfaction in Isolated Patient Care
Brief Title: The Effect of Standardised Patient Simulation in Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Hamiyet KIZIL, Assistant Professor, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-3
Record Dates: First submitted 2024-08-18; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Nursing Caries
Keywords: Care; isolation; nursing; simulation; standardised patient

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Training Group (Experimental): Students in the control group were taken to the laboratory practice within one week after the training presentation. Students were expected to act in accordance with the skills of isolation precautions in line with the 'Sample Scenario'. The individual in this scenario was an individual who was diagnosed with Covid-19 and suffered from anxiety due to isolation and neglected some rules. The performance of the students was evaluated with the Skill Evaluation Form for Isolated Patient Care. The students were asked to fill out the 'Satisfaction Survey on Training Methods' at the end of the application. Their opinions and suggestions regarding the training they attended were also taken.
  Interventions: Other: Control
- Training Group for Standardised Patient Simulation (Experimental): One week after the training presentation, the experimental group was invited to the simulation training. Simulation training was carried out in a hospital environment. Materials to be used in standardised patient and isolated patient care were made available in the room. The students were introduced to the field, scenario information on the subject and general principle frameworks. Students were included in groups in the simulation training created in line with the 'Simulation Scenario'. The scenario was prepared in line with the Healthcare Simulation Standards of Best PracticeTM of the International Nursing Association for Clinical Simulation and Learning (INACSL) standards (31) and submitted for expert opinion.
  Interventions: Other: Training Group for Standardised Patient Simulation

INTERVENTIONS:
Other: Control — Students in the control group were taken to the laboratory practice within one week after the training presentation. Students were expected to act in accordance with the skills of isolation precautions in line with the 'Sample Scenario'.
  Other Names: No intervention was performed
  Arms: Traditional Training Group
Other: Training Group for Standardised Patient Simulation — One week after the training presentation, the experimental group was invited to the simulation training. Simulation training was carried out in a hospital environment. Materials to be used in standardised patient and isolated patient care were made availa
  Other Names: Before the training, the students were introduced to the field, scenario information on the subject and general principle frameworks
  Arms: Training Group for Standardised Patient Simulation

SUMMARY:
With the coronavirus outbreak, the experience of nursing students with personal protective equipment is one of the issues of interest. The competence of nursing students is important in terms of the fact that outbreaks will persist in the future. In this study, the effect of standardised patient method in training of isolated patient care in terms of knowledge, skills and satisfaction of nursing students was investigated. A experimental design was employed in this study, involving a total of 80 nursing university students, with 40 participants in the experimental group and 40 in the control group. In the study, pre-test-post-test knowledge exam, isolated patient care skills and training satisfaction of nursing students were evaluated. In addition to descriptive statistical methods, chi-square, fisher exact and t-tests were used in the evaluation of the data.

DETAILED DESCRIPTION:
Material and method of the research:

Type of Study: The study was designed as randomized controlled experimental type.

Research Hypotheses Hypothesis 1 (H1): H1: The knowledge level of nursing students who received simulation training with standardised patient is higher in isolated patient care training.

Hypothesis 2 (H2): Nursing students who received simulation training with standardised patient have higher skill level in isolated patient care training.

Hypothesis 3 (H3): The satisfaction of nursing students who received simulation training with standardised patient is higher in isolated patient care training.

Population and Sample of the Study: The population of the study consisted of the senior students of a foundation university in Istanbul (N=110). The study was conducted in the spring term of the 2022-2023 academic year within the scope of the 'Nursing Principles' course. Power analysis was performed to determine the number of people to be included in the study. As a similar study in the related literature, Park & Kim (2020) calculated the effect size for the difference in knowledge level as 0.857 in the study (28). In order to exceed the 95% value in determining the power of the study, it was determined that 62 people (df=60; t=1.671), including 31 people in groups with a significance level of 5% and an effect size of 0.857, should be reached. Considering the high power of the test and the losses in the study, a total of 80 students (40 experimental; 40 control) were reached.

Data Collection Tools: The data were collected using "The Student Information Form", "Knowledge Test on Isolated Patient Care', "Skills Assessment Form for Isolated Patient Care" and "Satisfaction Survey on Training Methods".

Analysis of Data: The data obtained in the study were analysed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 software. Number, percentage, mean, standard deviation were used as descriptive statistical methods in the evaluation of the data. Kurtosis and Skewness values were analysed to determine whether the research variables were normally distributed. In the related literature, the results of kurtosis and skewness values of the variables between +1.5 and -1.5 (32), +2.0 and -2.0 (33) are accepted as normal distribution. It was determined that the variables were normally distributed. Differences between the rates of categorical variables in independent groups were analysed with Chi-Square and Fisher exact tests. T-test was used to compare quantitative continuous data between two independent groups. Dependent groups t-test was used for comparison of intra-group measurements.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages 18-30
* Agreeing to participate in the study
* Being able to participate in the training and its implementation

Exclusion Criteria:

* not between the ages 18-30
* Lack of consent to participate in the study
* Absence from education and practice during the study period
* Request to leave during the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Skill Evaluation Form for Isolated Patient Care | 2 months
  This form was developed in accordance with the isolation precautions guideline of the CDC. The form includes 20 skill steps to be completed regarding isolation precautions. The skills included communication, isolation measures and scenario-specific care steps. The range of points that can be obtained from the form is between 0-100.
Knowledge Test on Isolated Patient Care | 2 Months
  There are 20 questions in the form created by the researchers in line with the literature. The scope of the questions included communication with the patient, use of protective equipment, hand washing and care practices. The range of points that can be obtained from the form is between 0-100.

SECONDARY OUTCOMES:
Satisfaction Survey for Training Methods | 2 Months
  The satisfaction survey on Training Methods was developed by Gürpınar (Cronbach's alpha: 0.84) and used in his studies . The survey consists of 16 propositions. Each proposition is scored according to a 5-point Likert scale (1 - strongly disagree, 2 - disagree, 3 - undecided, 4 - agree, 5 - strongly agree). It was determined that the higher the mean score of the scale, the higher the students' satisfaction with the training method, and the lower the mean score of the scale, the lower their satisfaction with the training method. In the evaluation of the scale, students' satisfaction with the Training Methods is scored at least 16 and at most 80 points.

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Kızıl, PhD, Principal Investigator — Beykent University
Locations (1):
- Beykent Üniversity, Istanbul, Beykent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim E, Kim SS, Kim S. Effects of Infection Control Education for Nursing Students Using Standardized Patients vs. Peer Role-Play. Int J Environ Res Public Health. 2020 Dec 26;18(1):107. doi: 10.3390/ijerph18010107. PMID 33375222
- [Result] Bouget Mohammedi S, Landelle C. Review of literature: Knowledge and practice of standard precautions by nursing student and teaching techniques used in training. Am J Infect Control. 2023 May;51(5):574-581. doi: 10.1016/j.ajic.2022.08.032. Epub 2022 Sep 6. PMID 36075296